CLINICAL TRIAL: NCT04273165
Title: A Phase 2 Clinical Trial to Test the Safety and Efficacy of Etravirine in Friedreich Ataxia Patients
Brief Title: Safety and Efficacy of Etravirine in Friedreich Ataxia Patients
Acronym: FAEST1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002618-38; 2019-002618-38 (EudraCT Number)
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — etravirine

STUDY DESIGN:
Intervention Model Description: dose comparison in open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etravirine Dose 1 (Active Comparator): Etravirine dose 200 mg per diem(100+100)
  Interventions: Drug: Etravirine Tablets
- Etravirine Dose 2 (Active Comparator): Etravirine dose 400 mg per diem (200+200)
  Interventions: Drug: Etravirine Tablets

INTERVENTIONS:
Drug: Etravirine Tablets — Daily etravirine BID with 100 or 200 tablets for 4 months

SUMMARY:
A drug repositioning effort provided evidence supporting the possible use of Etravirine, a drug approved for the treatment of HIV infections in patients starting from 2 years of age, as a treatment for FA. We found that Etravirine is able to increase Frataxin protein both in vitro - in cells derived from FA patients - and in vivo - in the heart and skeletal muscle of Frataxin-deficient YG8 mice. Because of these findings, and since Etravirine displays a generally favorable safety profile, we plan to launch an open-label, phase 2 clinical trial aimed at assessing the safety and efficacy of Etravirine in FA patients. We aim at recruiting 30 FA patients. 15 will be treated with Etravirine for 4 months at 200 mcg/day and 15 will be treated with Etravirine for 4 months at 400 mg/day. Efficacy primary endpoint will be represented changes in peak VO2 as measured by incremental cycle ergometer exercise test. Secondary endpoints will include maximal workload, SARA score, cardiac measures, Frataxin protein levels in peripheral blood mononuclear cells and molecular analysis of Frataxin mRNA translation efficiency. Complete sets of data will be collected 4 months before the start of the treatment (T -4), at the start (T0), after 2 months (T2), at the end of the treatment (T4) and 4 months after the termination of the treatment (T8).

DETAILED DESCRIPTION:
Friedreich ataxia is a rare progressive neurodegenerative disease presenting in childhood or late adolescence for which no treatment is currently available. The disease is caused by the defective synthesis of Frataxin, a mitochondrial protein synthesized by the FXN gene. Over 95% of patients carry a homozygous intronic GAA expansion that impairs FXN gene transcription and translation. The persistence of an intact reading frame within the genome of most FRDA patients opens the way to treatment attempts that target FXN gene transcription and mRNA translation to increase endogenous Frataxin levels and balance the complex metabolic consequences of Frataxin deficiency. The disease is characterized by a relentless progression involving motor coordination (ataxia), heart function and structure (hypertrophic cardiopathy), exercise capacity (impaired bioenergetics with reduced aerobic capacity), endocrine function (diabetes) visual and auditory function (optic atrophy and hearing loss).

By screening a library of 853 FDA-approved drugs, we found a few drugs that are capable to upregulate Frataxin in vitro. Among them, we selected and focused on Etravirine for its generally favorable safety profile. In Friedreich ataxia (FRDA) patients-derived cells, we found that Etravirine upregulates mature Frataxin protein, enhances the activity of aconitase and confers resistance to oxidative stress. Etravirine appears to upregulate Frataxin protein by a mechanism of action involving the redistribution of frataxin mRNA on heavy polysomes and consequent enhancement of Frataxin mRNA translation. Moreover, in collaboration with Dr. Mark Pook, Brunel University, London, we obtained evidence that Etravirine is able to upregulate Frataxin protein in the heart and in the skeletal muscle of YG8 mice dosed orally for 5 days with Etravirine (unpublished).

Etravirine is a diarylpyrimidine that acts as a non-nucleoside reverse transcriptase inhibitor. It was approved in 2008 by the FDA (tradename Intelence) for the treatment of patients affected by HIV that are resistant to other drugs. In 2018 the label was extended to include patients 2 years of age and older. The FDA label reports no contraindications. Etravirine is administered orally in tablets.

Preliminary Results

In collaboration with Dr. Mark Pook, Brunel University, London, we tested whether Etravirine is able to upregulate Frataxin protein in tissues of YG8 mice. Five YG8 mice were dosed for 5 days orally with Etravirine (10 mg/Kg) and five YG8 mice were dosed for 5 days orally with vehicle. Four hrs after last dosing, all the mice were sacrificed and protein extracts prepared from tissues. SDS-PAGE followed by immunoblotting revealed that Frataxin protein was significantly increased in the heart and in the skeletal muscle of Etravirine-dosed mice, compared to vehicle-dosed mice.

Specific Aims

Because of its ability to upregulate Frataxin protein and rescue phenotypic defects in FA patient-derived cells and because of its safety and approved use in children, Etravirine represents an attractive potential therapeutic for FA. Aim of the study, therefore, will be assessing the safety and efficacy of Etravirine in a small population of young FA patients.

Experimental Plan Study design. The study will be a randomized open-label Phase 2 clinical trial, to investigate the safety and efficacy of Etravirine in FA patients.

Study population. We aim at enrolling 30 FA patients, aged 10 to 40 years over a period of 6 months. Enrollment will be done by advertising the study through the patients' associations and among FA patients currently followed at the Medea site (50 subjects at present time). The patients will be screened and evaluated in the tertiary care hospital setting where Dr Martinuzzi is active. Treatment will be carried on at home following the prescription given to the patients at each visit.

Study Intervention. Recruited subjects will be randomized 1:1 by a computer-generated randomization sequence to either of the two dose regimens: Etravirine orally 200 mg/day (100 mg cpr x 2, morning and evening) for 4 months or Etravirine 400 mg/day (one 200 mg cpr x 2 morning and evening) for 4 months. Treatment will start only after the 4 months pre-treatment period will be completed and after the T0 evaluation visit.

Withdrawal criteria. Failure to comply with the study follow-up visits or with the treatment protocol. Occurrence of a SUSAR (suspected unexpected severe adverse reaction) deemed related to the drug treatment.

Stopping rules. The entire study will be interrupted: 1) When the third SUSAR occurs in different patients. 2) On the occurrence of the same SUSAR in two different patients. 3) Upon the occurrence of the first serious adverse event judged to be related to the investigational drug, which has endangered a patient's life or caused permanent damage. 4) Upon the exclusion of the third patient from the trial.

Endpoints

1. Safety. Hematochemical parameters (Blood cell count, glycaemia, BUN, Creatinine, AST, ALT, yGT, ferritin, Troponine) will be acquired 4 months before the start of the Etravirine treatment (T -4), at the start of the treatment (T0), after 2 months (T2), at the end of the treatment (T4) and 4 months after the termination of the treatment (T8). A physical evaluation including vital parameters assessment and skin inspection for possible rash will be completed at enrollment and at each follow up visit. A detailed questionnaire listing all known adverse events associated with Etravirine will be distributed to all patients and reviewed at each follow up visit. Any additional AE will be registered irrespective of its likely connection with the treatment.
2. Efficacy Primary endpoint. Primary endpoint of the study will be the change in peak aerobic capacity (VO2 peak) achieved by participants during a standardized incremental exercise test by cycle ergometer. Peak VO2 normalized by weight, is a very stable objective measure of aerobic capacity. FA is associated with significant decrease (50-60% less) aerobic fitness as measured by standardized exercise testing and its measure has been employed as primary end point in FA intervention trials several times.

Secondary endpoints. Secondary endpoints will include:

* clinical measures of the disease as quantitated by the Scale for the assessment and Rating of Ataxia (SARA); SARA is the most sensitive functional composite measure of performance developed specifically for ataxic disorders;
* Critical cardiac parameters (including interventricular septal wall thickness, left ventricular wall thickness, left ventricular ejection fraction, Sokolow-Lyon index); Heart is primarily affected in FA showing progressive mostly left ventricular hypertrophic. Cardiomyopathy is the main determinant of survival in this population. The ECG changes summarized by the Sokolow-Lyon index (∆%QRS-voltage) are reliable indicators of ventricular hypertrophy. Echocardiography can detect and measure very precisely the extent and severity of heart hypertrophic changes;
* Additional exercise indicators: maximal workload (W/Kg) reached at exhaustion during the incremental exercise test;
* WHO-DAS 2.0 is an internationally validated widely applied disease non-specific measure of disability developed by WHO within the framework of the biopsychosocial model of functioning and disability. It asks the subject to score in terms of severity and duration any difficulty experienced in the 30 previous days in 6 main life areas. The interview format will be used and the results will be computed as normalized scores. This measure has been validated only above age 16 and thus will be administered only to subjects >16 years of age.
* Frataxin protein levels as measured in peripheral blood cells. Frataxin protein will be quantitated by SDS-PAGE and immunoblotting in protein extracts from peripheral blood mononuclear cells. At the same time points, to assess the effect of Etravirine on Frataxin mRNA translation, the distribution of Frataxin mRNA in the translationally active heavy polysomal fraction, will be determined in extracts from peripheral blood mononuclear cells.

Sample size calculation. Sample size was calculated considering the primary endpoint. VO2 at peak in controls subjects shows a value >16.2 with a test-retest variability of ± 4 ml/min/Kg. Workload at peak is expected to be >3W/Kg in control subjects with a SD of ± 0.8. This parameter is reduced by approximately 50% in FA patients with similar SD values. Considering an alpha error of 0.05 and a statistical power of 80%, the needed number of participants is 30.

Statistical analysis. Both primary and secondary endpoints will be analyzed using multivariate linear mixed models modeling timepoints as a repeated within-subject factor. Mixed models have the advantage of being able to account for heterogeneous distances between timepoints, missing data as well as unequal variances and covariances. In order to account for possible confounds due to inter-patient variability, all models will include sex, age at onset, disease duration, years of education and number of GAA1 repeats within the smaller FXN allele as covariates of no interest. When a statistically significant (p<0.05) overall effect of time is found, pairwise comparisons between timepoints were will be performed and corrected for multiple comparisons across pairs of timepoints using the Dunn-Šidák correction.

ELIGIBILITY:
Inclusion Criteria:

* Molecularly defined FA diagnosis (at least one expanded FXN allele),
* ability to complete maximal exercise testing (being able to ride a recumbent exercise ergometer at 60 rpm with no added resistance for at least 3 minutes),
* willingness to participate, as shown by the signed consent form.

Exclusion Criteria:

* Known intolerance to any of the components of the drug preparation.
* Ongoing treatment with Etravirine or other experimental therapeutics under study for FA (e.g. IFNy, erythropoietin, nicotinamide, etc.).
* Previous treatment, if any, should have been stopped at least 4 weeks before study entry.
* Severe medical condition likely to interfere with drug absorbance and distribution (liver or kidney failure, severe metabolic unbalance), significant cardiac disease

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Adverse event number and severity | 4 months
  description and count of AE and SAE to document the safety of etravirine treatment at 200 mg/die and 400mg/die in FA patients

SECONDARY OUTCOMES:
VO2 max increase | 12 months
  efficacy of etravirine treatment in increasing aerobic capacity in FA patients comparing pre and post treatment periods

OTHER OUTCOMES:
Scale for the Assessment and Rating of Ataxia | 12 months
  Scale for the Assessment and Rating of Ataxia (SARA) score change comparing pre-, during- and post- treatment evaluations. SARA scores ataxia on a 0-40 points scale where 0 means no ataxia and 40 most severe ataxia
Cardiac wall thickness (in mm) | 12 months
  cardiac wall thickness (in mm) as measured by standard Echo cardiography
Frataxin measurement | 12 months
  Frataxin protein content in peripheral blood mononuclear cells
short form 36 scale for quality of life | 12 months
  changes in QoL as measured by the short form 36 (SF36) scale and disability as measured with the World Health Organization Disability Assessment schedule 2.0 (WHO-DAS 2.0) during the study period. Both tools are graded on a 0-100 scale where 100 is best and 0 is worst.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea Scientific Institute, Pieve di Soligo Research Centre, Pieve di Soligo, TV, Italy

REFERENCES:
- [Background] Paparella G, Straga C, Pesenti N, Dal Molin V, Martorel GA, Merotto V, Genova C, Piazza A, Piccoli G, Panzeri E, Rufini A, Testi R, Martinuzzi A. A Pilot Phase 2 Randomized Trial to Evaluate the Safety and Potential Efficacy of Etravirine in Friedreich Ataxia Patients. Children (Basel). 2024 Aug 9;11(8):958. doi: 10.3390/children11080958. PMID 39201893
- [Background] Alfedi G, Luffarelli R, Condo I, Pedini G, Mannucci L, Massaro DS, Benini M, Toschi N, Alaimo G, Panarello L, Pacini L, Fortuni S, Serio D, Malisan F, Testi R, Rufini A. Drug repositioning screening identifies etravirine as a potential therapeutic for friedreich's ataxia. Mov Disord. 2019 Mar;34(3):323-334. doi: 10.1002/mds.27604. Epub 2019 Jan 9. PMID 30624801